CLINICAL TRIAL: NCT07356440
Title: Effect of Consumption of Vegetable Protein-enriched Biscuits and Vitamin D Supplementation on the Progression of Sarcopenia in Elderly Subjects
Brief Title: Effect of the Consumption of Cookies Enriched With Plant Proteins and of a Vitamin D Supplement on the Progression of Sarcopenia in the Elderly
Acronym: SARC-PEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Udine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEUR-2024-Sper-39
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia in Elderly; Sarcopenia; Nutritional Intervention; Microbiome Analysis; Muscle Mass and Strength; Biomarkers / Blood; Quality of Life Outcomes
Keywords: sarcopenia; elderly; pea proteins; vitamin D; snack
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-enriched biscuit + Vitamin D3 (Experimental): Participants will consume daily one portion (50 g) of experimental biscuits made with wheat flour and pea protein hydrolysate, and take 4 drops of vitamin D3 supplement in extra virgin olive oil.
  Interventions: Dietary Supplement: Vitamin D3 supplement; Other: Protein-enriched biscuits
- Control Biscuit + Placebo Oil (Placebo Comparator): Participants will consume daily one portion (50 g) of control biscuits (same recipe without pea protein hydrolysate), and take 4 drops of placebo oil (extra virgin olive oil without vitamin D3).
  Interventions: Other: Control biscuit; Other: Placebo oil

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplement — Four daily drops of vitamin D3 dissolved in extra virgin olive oil. Used in the Experimental Arm.
  Arms: Protein-enriched biscuit + Vitamin D3
Other: Protein-enriched biscuits — Daily portion (50 g) of biscuits made with wheat flour and pea protein hydrolysate. Used in the Experimental Arm.
  Arms: Protein-enriched biscuit + Vitamin D3
Other: Control biscuit — Daily portion (50 g) of control biscuits made with wheat flour, without pea protein hydrolysate.
  Arms: Control Biscuit + Placebo Oil
Other: Placebo oil — Four daily drops of placebo oil (extra virgin olive oil without vitamin D3).
  Arms: Control Biscuit + Placebo Oil

SUMMARY:
The ageing population makes it necessary to find effective strategies for the prevention of sarcopenia (the progressive loss of muscle mass and strength and a decline in physical performance) that can be counteracted with foods containing protein and adequate intake of vitamin D. This study will evaluate the effectiveness of consuming a food based on plant proteins and vitamin D supplementation. Intervention studies in humans conducted to date have mostly focused on the effect of animal proteins (mainly from whey) on disease progression. A study on the effect of pea proteins has not yet been conducted and will provide information on the effectiveness of these proteins in modulating markers linked to the disease. The effect on the gut microbiota will also be considered, as the existence of a gut-muscle axis has been suggested, in which microbial genera producing short-chain fatty acids have been linked to a positive effect on muscle mass through anabolic stimulation. Thus, the analysis of the modulation of the intestinal microbiota, through the dietary intervention proposed in this study, may represent a further step in research related to the prevention of this disease. Sarcopenic volunteers aged between 65 and 75 will be recruited to consume either a shortbread biscuit made with wheat flour enriched with hydrolysed pea protein and a vitamin D supplement in extra virgin olive oil, or a control biscuit and a placebo (extra virgin olive oil) for 12 weeks. The study will be randomised, parallel, single-blind. The effect of consuming the experimental biscuit and vitamin D supplementation compared to that of a traditional control biscuit and a placebo oil solution will be evaluated on certain markers related to sarcopenia. In particular, the following will be considered: muscle strength, measuring grip strength and leg strength (chair stand test); muscle mass through the measurement of appendicular muscle mass, and the calculation of the appendicular muscle mass index; physical performance using the Short Physical Performance Battery; the inflammatory response and other blood biomarkers related to sarcopenia. In addition, the following will be assessed: dietary habits through a food diary and quality of life through the SarQoL questionnaire. Finally, the effect of nutritional intervention on the modulation of the gut microbiota will be evaluated through 16S rRNA sequencing and bioinformatic analysis of the data.

DETAILED DESCRIPTION:
Sarcopenia, characterized by the age-related loss of muscle mass, strength, and physical performance, is a growing public health concern given the global aging population. Nutritional interventions, particularly those involving protein and vitamin D supplementation, have shown promise in managing sarcopenia. However, physical activity-the standard treatment-is often not feasible for frail or bedridden elderly individuals, highlighting the need for alternative strategies.

This randomized, single-blind, parallel-design clinical trial aims to evaluate the effect of consuming a shortbread biscuit enriched with hydrolyzed pea protein, combined with a daily dose of vitamin D3 (800 IU/day), on muscle mass, muscle strength, physical performance, and gut microbiota composition in sarcopenic individuals aged 65-75 years. The study will enroll 74 participants meeting specific inclusion criteria (e.g., low appendicular skeletal muscle mass index, poor SPPB score, and sufficient cognitive and nutritional status).

Participants will be randomly assigned to one of two groups:

1. Intervention Group: Receives a 50 g daily portion of a functional biscuit enriched with hydrolyzed pea protein, and 4 drops/day of a vitamin D3 supplement (providing 20 μg/day).
2. Control Group: Receives a similar biscuit without added protein and a placebo oil (extra virgin olive oil) in place of vitamin D3.

The intervention will last for 12 weeks. Measurements will be taken at baseline, mid-point (6 weeks), and study end (12 weeks), including handgrip strength, chair stand test, bioimpedance-based muscle mass, and SPPB. Blood samples will be analyzed for markers related to inflammation (e.g., CRP, IL-6, TNF-α), oxidative stress (oxLDL), anabolic signaling (IGF-1), and vitamin D status (25-hydroxycholecalciferol), among others. Gut microbiota composition and short-chain fatty acid (SCFA) production will be assessed via stool sample analysis and 16S rRNA sequencing.

Participants will also complete quality-of-life (SarQoL) and food frequency questionnaires, along with 3-day dietary diaries at each time point. Compliance will be monitored via diary entries and return of supplement containers. A sample size of 74 participants (32 per group + 15% dropout) was calculated to detect a 25% difference in treatment success (as defined by surpassing the sarcopenia threshold in ASMI).

The study further investigates the potential of plant-based protein sources, particularly hydrolyzed pea protein, to serve as effective dietary interventions in the elderly. It also explores the gut-muscle axis, examining how nutritional modulation of the microbiota may impact sarcopenia-related outcomes.

The trial is conducted at the Internal Medicine Unit 2 of the S. Maria della Misericordia Hospital (Udine, Italy) under the coordination of Prof. Alessandro Cavarape. All procedures follow ethical guidelines and include appropriate monitoring for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Ishii equation values: patients with a score ≥105 for males and ≥120 for females will be included. The Ishii screening test is a widely used method that estimates the probability of sarcopenia using a score derived from an equation based on three variables: age, grip strength, and calf circumference.
* Appendicular skeletal muscle mass index (ASMI): <7.0 kg/m2 for males and <5.5 kg/m2 for females.
* Short physical performance battery score ≤8
* Body mass index ≥19 <30 kg/m2
* Ability to act

Exclusion Criteria:

* Body mass index <19≥30 kg/m2
* Diagnosis of cancer in the previous five years;
* Regular intake of vitamin D supplements;
* Dysphagia and difficulty chewing;
* Allergy or other intolerances to gluten;
* Allergy to eggs;
* Intestinal disorders (Crohn's disease, ulcerative colitis, bacterial contamination syndrome, constipation, coeliac disease, irritable bowel syndrome) that could have an impact on the intestinal microbiota;
* Pacemaker wearers;
* Acute inflammation (CRP >10 mg/L);
* Anaemia (haemoglobin <13 g/dL in men; <12 g/dL women);
* Renal failure (glomerular filtration rate (GFR) >45 mL/min/1.73 m2);
* Chronic liver disease (transaminases < 40 IU/L men, < 35 IU/L women);
* Inability to act

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Appendicular Skeletal Muscle Index (ASMI) | Enrollment, baseline, week 6 and week 12 (end of the treatment)
  ASMI will be calculated by dividing appendicular skeletal muscle mass (measured by bioelectrical impedance analysis, BIA 101; BIVA® PRO, Akern Srl, Pisa, Italia) by height squared (kg/m²).

SECONDARY OUTCOMES:
Muscle strenght | Baseline, week 6 and week 12 (end of the treatment)
  The muscle strenght will be measured using two different analysis Handgrip Strength: Measured using Electronic Hand Dynamometer EH101, dominant hand, two attempts.
  Chair Stand Test: Number of stands in 30 seconds without upper limb support.
Physical performance (SPPB score) | Enrollment, baseline, week 6 and week 12 (end of the treatment)
  Short Physical Performance Battery (balance tests, 4-meter walk, 5 sit-to-stand repetitions).
Blood biomarkers | Baseline, week 6 and week 12 (end of the treatment)
  Plasma levels of PCR, IL-6, TNF-α, oxLDL, IGF-1, 25-hydroxyvitamin D, albumin, triglycerides, leptin, and C-terminal agrin fragment.
Gut micorbiome modulation and metabolites | Baseline at at week 12 (end of the treatment)
  Analysis of fecal samples for SCFA production (via gas chromatography) and microbiota composition (16S sequencing, α-diversity, relative abundance of sarcopenia-associated genera: Roseburia, Eubacterium, Lachnospira, Ruminococcus).
Nutritional intake | Baseline, week 6 and week 12 (end of the treatment)
  3-day dietary records
Nutritional habits | Enrollment
  food frequency questionnaire (FFQ).
Quality of life of sarcopenic patients | Baseline, week 6 and week 12 (end of the treatment)
  SarQoL questionnaire to assess health-related quality of life in sarcopenic subjects
SARC-F | At the screening
  Screening tool that can be rapidly implemented by clinicians to identify probable sarcopenic patients.
Mini Nutritional Assessment (MNA®) | At the screening
  The MNA® is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition.
Mini Mental State Examination (MMSE) | At the screening
  It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Cavarape, M.D., Principal Investigator — Azienda Sanitaria Universitaria del Friuli Centrale (ASU FC)
Locations (3):
- Italy (3):
  - Department of Agricultural, Food, Environmental and Animal Sciences, Udine, Udine
  - Laboratory of Immunology, Department of Medicine, Udine, Udine
  - Outpatient Clinic of Internal Medicine 2, Central Friuli University Health Authority (ASU FC), Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akune T, Muraki S, Oka H, Tanaka S, Kawaguchi H, Tokimura F, Yoshida H, Suzuki T, Nakamura K, Yoshimura N. Incidence of certified need of care in the long-term care insurance system and its risk factors in the elderly of Japanese population-based cohorts: the ROAD study. Geriatr Gerontol Int. 2014 Jul;14(3):695-701. doi: 10.1111/ggi.12155. Epub 2013 Sep 11. PMID 24020635
- [Background] Anagnostis P, Dimopoulou C, Karras S, Lambrinoudaki I, Goulis DG. Sarcopenia in post-menopausal women: Is there any role for vitamin D? Maturitas. 2015 Sep;82(1):56-64. doi: 10.1016/j.maturitas.2015.03.014. Epub 2015 Mar 27. PMID 25882761
- [Background] Bauer J, Biolo G, Cederholm T, Cesari M, Cruz-Jentoft AJ, Morley JE, Phillips S, Sieber C, Stehle P, Teta D, Visvanathan R, Volpi E, Boirie Y. Evidence-based recommendations for optimal dietary protein intake in older people: a position paper from the PROT-AGE Study Group. J Am Med Dir Assoc. 2013 Aug;14(8):542-59. doi: 10.1016/j.jamda.2013.05.021. Epub 2013 Jul 16. PMID 23867520
- [Background] Beasley JM, Wertheim BC, LaCroix AZ, Prentice RL, Neuhouser ML, Tinker LF, Kritchevsky S, Shikany JM, Eaton C, Chen Z, Thomson CA. Biomarker-calibrated protein intake and physical function in the Women's Health Initiative. J Am Geriatr Soc. 2013 Nov;61(11):1863-71. doi: 10.1111/jgs.12503. Epub 2013 Oct 28. PMID 24219187
- [Background] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Dardenne N, Bruyere O. Validation of the SarQoL(R), a specific health-related quality of life questionnaire for Sarcopenia. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):238-244. doi: 10.1002/jcsm.12149. Epub 2016 Oct 22. PMID 27897430
- [Background] Behrouzi P, Grootswagers P, Keizer PLC, Smeets ETHC, Feskens EJM, de Groot LCPGM, van Eeuwijk FA. Dietary Intakes of Vegetable Protein, Folate, and Vitamins B-6 and B-12 Are Partially Correlated with Physical Functioning of Dutch Older Adults Using Copula Graphical Models. J Nutr. 2020 Mar 1;150(3):634-643. doi: 10.1093/jn/nxz269. PMID 31858107
- [Background] Bischoff-Ferrari HA, Orav JE, Kanis JA, Rizzoli R, Schlogl M, Staehelin HB, Willett WC, Dawson-Hughes B. Comparative performance of current definitions of sarcopenia against the prospective incidence of falls among community-dwelling seniors age 65 and older. Osteoporos Int. 2015 Dec;26(12):2793-802. doi: 10.1007/s00198-015-3194-y. Epub 2015 Jun 12. PMID 26068298
- [Background] Boutry-Regard C, Vinyes-Pares G, Breuille D, Moritani T. Supplementation with Whey Protein, Omega-3 Fatty Acids and Polyphenols Combined with Electrical Muscle Stimulation Increases Muscle Strength in Elderly Adults with Limited Mobility: A Randomized Controlled Trial. Nutrients. 2020 Jun 23;12(6):1866. doi: 10.3390/nu12061866. PMID 32585837
- [Background] Bradlee ML, Mustafa J, Singer MR, Moore LL. High-Protein Foods and Physical Activity Protect Against Age-Related Muscle Loss and Functional Decline. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):88-94. doi: 10.1093/gerona/glx070. PMID 28549098
- [Background] Chanet A, Verlaan S, Salles J, Giraudet C, Patrac V, Pidou V, Pouyet C, Hafnaoui N, Blot A, Cano N, Farigon N, Bongers A, Jourdan M, Luiking Y, Walrand S, Boirie Y. Supplementing Breakfast with a Vitamin D and Leucine-Enriched Whey Protein Medical Nutrition Drink Enhances Postprandial Muscle Protein Synthesis and Muscle Mass in Healthy Older Men. J Nutr. 2017 Dec;147(12):2262-2271. doi: 10.3945/jn.117.252510. Epub 2017 Aug 23. PMID 28835387
- [Background] Chang SS, Chen LH, Huang KC, Huang SW, Chang CC, Liao KW, Hu EC, Chen YP, Chen YW, Hsu PC, Huang HY. Plant-based polyphenol rich protein supplementation attenuated skeletal muscle loss and lowered the LDL level via gut microbiota remodeling in Taiwan's community-dwelling elderly. Food Funct. 2023 Oct 16;14(20):9407-9418. doi: 10.1039/d3fo02766j. PMID 37795525
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cho MR, Lee S, Song SK. A Review of Sarcopenia Pathophysiology, Diagnosis, Treatment and Future Direction. J Korean Med Sci. 2022 May 9;37(18):e146. doi: 10.3346/jkms.2022.37.e146. PMID 35535373
- [Background] Coelho-Junior HJ, Calvani R, Goncalves IO, Rodrigues B, Picca A, Landi F, Bernabei R, Uchida MC, Marzetti E. High relative consumption of vegetable protein is associated with faster walking speed in well-functioning older adults. Aging Clin Exp Res. 2019 Jun;31(6):837-844. doi: 10.1007/s40520-019-01216-4. Epub 2019 May 21. PMID 31115875
- [Background] Cox NJ, Bowyer RCE, Ni Lochlainn M, Wells PM, Roberts HC, Steves CJ. The composition of the gut microbiome differs among community dwelling older people with good and poor appetite. J Cachexia Sarcopenia Muscle. 2021 Apr;12(2):368-377. doi: 10.1002/jcsm.12683. Epub 2021 Feb 13. PMID 33580637
- [Background] Sura L, Madhavan A, Carnaby G, Crary MA. Dysphagia in the elderly: management and nutritional considerations. Clin Interv Aging. 2012;7:287-98. doi: 10.2147/CIA.S23404. Epub 2012 Jul 30. PMID 22956864
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] De Buyser SL, Petrovic M, Taes YE, Toye KR, Kaufman JM, Lapauw B, Goemaere S. Validation of the FNIH sarcopenia criteria and SOF frailty index as predictors of long-term mortality in ambulatory older men. Age Ageing. 2016 Sep;45(5):602-8. doi: 10.1093/ageing/afw071. Epub 2016 Apr 28. PMID 27126327
- [Background] Decarli A, Franceschi S, Ferraroni M, Gnagnarella P, Parpinel MT, La Vecchia C, Negri E, Salvini S, Falcini F, Giacosa A. Validation of a food-frequency questionnaire to assess dietary intakes in cancer studies in Italy. Results for specific nutrients. Ann Epidemiol. 1996 Mar;6(2):110-8. doi: 10.1016/1047-2797(95)00129-8. PMID 8775590
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820
- [Background] Dos Santos L, Cyrino ES, Antunes M, Santos DA, Sardinha LB. Sarcopenia and physical independence in older adults: the independent and synergic role of muscle mass and muscle function. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):245-250. doi: 10.1002/jcsm.12160. Epub 2016 Nov 8. PMID 27897417
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Ganapathy A, Nieves JW. Nutrition and Sarcopenia-What Do We Know? Nutrients. 2020 Jun 11;12(6):1755. doi: 10.3390/nu12061755. PMID 32545408
- [Background] Gazzani D, Zamboni F, Spelta F, Ferrari P, Mattioli V, Cazzoletti L, Zanolin E, Tardivo S, Ferrari M. Vegetable but not animal protein intake is associated to a better physical performance: a study on a general population sample of adults. Food Nutr Res. 2019 Sep 19;63. doi: 10.29219/fnr.v63.3422. eCollection 2019. PMID 31565042
- [Background] Gorissen SHM, Witard OC. Characterising the muscle anabolic potential of dairy, meat and plant-based protein sources in older adults. Proc Nutr Soc. 2018 Feb;77(1):20-31. doi: 10.1017/S002966511700194X. Epub 2017 Aug 29. PMID 28847314
- [Background] Hawley-Hague H, Horne M, Campbell M, Demack S, Skelton DA, Todd C. Multiple levels of influence on older adults' attendance and adherence to community exercise classes. Gerontologist. 2014 Aug;54(4):599-610. doi: 10.1093/geront/gnt075. Epub 2013 Jul 30. PMID 23899623
- [Background] Herrera-Martinez AD, Munoz Jimenez C, Lopez Aguilera J, Crespin MC, Manzano Garcia G, Galvez Moreno MA, Calanas Continente A, Molina Puerta MJ. Mediterranean Diet, Vitamin D, and Hypercaloric, Hyperproteic Oral Supplements for Treating Sarcopenia in Patients with Heart Failure-A Randomized Clinical Trial. Nutrients. 2023 Dec 28;16(1):110. doi: 10.3390/nu16010110. PMID 38201939
- [Background] Huang RY, Yang KC, Chang HH, Lee LT, Lu CW, Huang KC. The Association between Total Protein and Vegetable Protein Intake and Low Muscle Mass among the Community-Dwelling Elderly Population in Northern Taiwan. Nutrients. 2016 Jun 17;8(6):373. doi: 10.3390/nu8060373. PMID 27322317
- [Background] Ishii S, Tanaka T, Shibasaki K, Ouchi Y, Kikutani T, Higashiguchi T, Obuchi SP, Ishikawa-Takata K, Hirano H, Kawai H, Tsuji T, Iijima K. Development of a simple screening test for sarcopenia in older adults. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:93-101. doi: 10.1111/ggi.12197. PMID 24450566
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Kang L, Li P, Wang D, Wang T, Hao D, Qu X. Alterations in intestinal microbiota diversity, composition, and function in patients with sarcopenia. Sci Rep. 2021 Feb 25;11(1):4628. doi: 10.1038/s41598-021-84031-0. PMID 33633246
- [Background] Kim MK, Baek KH, Song KH, Il Kang M, Park CY, Lee WY, Oh KW. Vitamin D deficiency is associated with sarcopenia in older Koreans, regardless of obesity: the Fourth Korea National Health and Nutrition Examination Surveys (KNHANES IV) 2009. J Clin Endocrinol Metab. 2011 Oct;96(10):3250-6. doi: 10.1210/jc.2011-1602. Epub 2011 Aug 10. PMID 21832109
- [Background] Lahiri S, Kim H, Garcia-Perez I, Reza MM, Martin KA, Kundu P, Cox LM, Selkrig J, Posma JM, Zhang H, Padmanabhan P, Moret C, Gulyas B, Blaser MJ, Auwerx J, Holmes E, Nicholson J, Wahli W, Pettersson S. The gut microbiota influences skeletal muscle mass and function in mice. Sci Transl Med. 2019 Jul 24;11(502):eaan5662. doi: 10.1126/scitranslmed.aan5662. PMID 31341063
- [Background] Leonel AJ, Alvarez-Leite JI. Butyrate: implications for intestinal function. Curr Opin Clin Nutr Metab Care. 2012 Sep;15(5):474-9. doi: 10.1097/MCO.0b013e32835665fa. PMID 22797568
- [Background] Liberman K, Njemini R, Luiking Y, Forti LN, Verlaan S, Bauer JM, Memelink R, Brandt K, Donini LM, Maggio M, Mets T, Wijers SLJ, Sieber C, Cederholm T, Bautmans I. Thirteen weeks of supplementation of vitamin D and leucine-enriched whey protein nutritional supplement attenuates chronic low-grade inflammation in sarcopenic older adults: the PROVIDE study. Aging Clin Exp Res. 2019 Jun;31(6):845-854. doi: 10.1007/s40520-019-01208-4. Epub 2019 May 2. PMID 31049877
- [Background] Lo JH, U KP, Yiu T, Ong MT, Lee WY. Sarcopenia: Current treatments and new regenerative therapeutic approaches. J Orthop Translat. 2020 Apr 30;23:38-52. doi: 10.1016/j.jot.2020.04.002. eCollection 2020 Jul. PMID 32489859
- [Background] Lu ZX, He JF, Zhang YC, Bing DJ. Composition, physicochemical properties of pea protein and its application in functional foods. Crit Rev Food Sci Nutr. 2020;60(15):2593-2605. doi: 10.1080/10408398.2019.1651248. Epub 2019 Aug 20. PMID 31429319
- [Background] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316
- [Background] McKendry J, Lowisz CV, Nanthakumar A, MacDonald M, Lim C, Currier BS, Phillips SM. The effects of whey, pea, and collagen protein supplementation beyond the recommended dietary allowance on integrated myofibrillar protein synthetic rates in older males: a randomized controlled trial. Am J Clin Nutr. 2024 Jul;120(1):34-46. doi: 10.1016/j.ajcnut.2024.05.009. Epub 2024 May 16. PMID 38762187
- [Background] Mesinovic J, Zengin A, De Courten B, Ebeling PR, Scott D. Sarcopenia and type 2 diabetes mellitus: a bidirectional relationship. Diabetes Metab Syndr Obes. 2019 Jul 8;12:1057-1072. doi: 10.2147/DMSO.S186600. eCollection 2019. PMID 31372016
- [Background] Milanovic Z, Pantelic S, Trajkovic N, Sporis G, Kostic R, James N. Age-related decrease in physical activity and functional fitness among elderly men and women. Clin Interv Aging. 2013;8:549-56. doi: 10.2147/CIA.S44112. Epub 2013 May 21. PMID 23723694
- [Background] Mioche L, Bourdiol P, Monier S, Martin JF, Cormier D. Changes in jaw muscles activity with age: effects on food bolus properties. Physiol Behav. 2004 Sep 30;82(4):621-7. doi: 10.1016/j.physbeh.2004.05.012. PMID 15327909
- [Background] Montiel-Rojas D, Nilsson A, Santoro A, Bazzocchi A, de Groot LCPGM, Feskens EJM, Berendsen AAM, Madej D, Kaluza J, Pietruszka B, Jennings A, Fairweather-Tait S, Battista G, Capri M, Franceschi C, Kadi F. Fighting Sarcopenia in Ageing European Adults: The Importance of the Amount and Source of Dietary Proteins. Nutrients. 2020 Nov 24;12(12):3601. doi: 10.3390/nu12123601. PMID 33255223
- [Background] Mori H, Tokuda Y. De-Training Effects Following Leucine-Enriched Whey Protein Supplementation and Resistance Training in Older Adults with Sarcopenia: A Randomized Controlled Trial with 24 Weeks of Follow-Up. J Nutr Health Aging. 2022;26(11):994-1002. doi: 10.1007/s12603-022-1853-1. PMID 36437767
- [Background] Morley JE, Abbatecola AM, Argiles JM, Baracos V, Bauer J, Bhasin S, Cederholm T, Coats AJ, Cummings SR, Evans WJ, Fearon K, Ferrucci L, Fielding RA, Guralnik JM, Harris TB, Inui A, Kalantar-Zadeh K, Kirwan BA, Mantovani G, Muscaritoli M, Newman AB, Rossi-Fanelli F, Rosano GM, Roubenoff R, Schambelan M, Sokol GH, Storer TW, Vellas B, von Haehling S, Yeh SS, Anker SD; Society on Sarcopenia, Cachexia and Wasting Disorders Trialist Workshop. Sarcopenia with limited mobility: an international consensus. J Am Med Dir Assoc. 2011 Jul;12(6):403-9. doi: 10.1016/j.jamda.2011.04.014. PMID 21640657
- [Background] Morley JE, Argiles JM, Evans WJ, Bhasin S, Cella D, Deutz NE, Doehner W, Fearon KC, Ferrucci L, Hellerstein MK, Kalantar-Zadeh K, Lochs H, MacDonald N, Mulligan K, Muscaritoli M, Ponikowski P, Posthauer ME, Rossi Fanelli F, Schambelan M, Schols AM, Schuster MW, Anker SD; Society for Sarcopenia, Cachexia, and Wasting Disease. Nutritional recommendations for the management of sarcopenia. J Am Med Dir Assoc. 2010 Jul;11(6):391-6. doi: 10.1016/j.jamda.2010.04.014. PMID 20627179
- [Background] Muir SW, Montero-Odasso M. Effect of vitamin D supplementation on muscle strength, gait and balance in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2011 Dec;59(12):2291-300. doi: 10.1111/j.1532-5415.2011.03733.x. PMID 22188076
- [Background] Ni Lochlainn M, Bowyer RCE, Moll JM, Garcia MP, Wadge S, Baleanu AF, Nessa A, Sheedy A, Akdag G, Hart D, Raffaele G, Seed PT, Murphy C, Harridge SDR, Welch AA, Greig C, Whelan K, Steves CJ. Effect of gut microbiome modulation on muscle function and cognition: the PROMOTe randomised controlled trial. Nat Commun. 2024 Feb 29;15(1):1859. doi: 10.1038/s41467-024-46116-y. PMID 38424099
- [Background] Picca A, Fanelli F, Calvani R, Mule G, Pesce V, Sisto A, Pantanelli C, Bernabei R, Landi F, Marzetti E. Gut Dysbiosis and Muscle Aging: Searching for Novel Targets against Sarcopenia. Mediators Inflamm. 2018 Jan 30;2018:7026198. doi: 10.1155/2018/7026198. eCollection 2018. PMID 29686533
- [Background] Piccirillo JF, Vlahiotis A, Barrett LB, Flood KL, Spitznagel EL, Steyerberg EW. The changing prevalence of comorbidity across the age spectrum. Crit Rev Oncol Hematol. 2008 Aug;67(2):124-32. doi: 10.1016/j.critrevonc.2008.01.013. Epub 2008 Mar 28. PMID 18375141
- [Background] Prokopidis K, Cervo MM, Gandham A, Scott D. Impact of Protein Intake in Older Adults with Sarcopenia and Obesity: A Gut Microbiota Perspective. Nutrients. 2020 Jul 30;12(8):2285. doi: 10.3390/nu12082285. PMID 32751533
- [Background] Reid-McCann RJ, Brennan SF, McKinley MC, McEvoy CT. The effect of animal versus plant protein on muscle mass, muscle strength, physical performance and sarcopenia in adults: protocol for a systematic review. Syst Rev. 2022 Apr 13;11(1):64. doi: 10.1186/s13643-022-01951-2. PMID 35418173
- [Background] Rondanelli M, Gasparri C, Barrile GC, Battaglia S, Cavioni A, Giusti R, Mansueto F, Moroni A, Nannipieri F, Patelli Z, Razza C, Tartara A, Perna S. Effectiveness of a Novel Food Composed of Leucine, Omega-3 Fatty Acids and Probiotic Lactobacillus paracasei PS23 for the Treatment of Sarcopenia in Elderly Subjects: A 2-Month Randomized Double-Blind Placebo-Controlled Trial. Nutrients. 2022 Oct 30;14(21):4566. doi: 10.3390/nu14214566. PMID 36364828
- [Background] Valenzuela RE, Ponce JA, Morales-Figueroa GG, Muro KA, Carreon VR, Aleman-Mateo H. Insufficient amounts and inadequate distribution of dietary protein intake in apparently healthy older adults in a developing country: implications for dietary strategies to prevent sarcopenia. Clin Interv Aging. 2013;8:1143-8. doi: 10.2147/CIA.S49810. Epub 2013 Sep 2. PMID 24039411
- [Background] Schaap LA, van Schoor NM, Lips P, Visser M. Associations of Sarcopenia Definitions, and Their Components, With the Incidence of Recurrent Falling and Fractures: The Longitudinal Aging Study Amsterdam. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1199-1204. doi: 10.1093/gerona/glx245. PMID 29300839
- [Background] Scott D, Blizzard L, Fell J, Giles G, Jones G. Associations between dietary nutrient intake and muscle mass and strength in community-dwelling older adults: the Tasmanian Older Adult Cohort Study. J Am Geriatr Soc. 2010 Nov;58(11):2129-34. doi: 10.1111/j.1532-5415.2010.03147.x. PMID 21054294
- [Background] Steffl M, Bohannon RW, Sontakova L, Tufano JJ, Shiells K, Holmerova I. Relationship between sarcopenia and physical activity in older people: a systematic review and meta-analysis. Clin Interv Aging. 2017 May 17;12:835-845. doi: 10.2147/CIA.S132940. eCollection 2017. PMID 28553092
- [Background] So D, Whelan K, Rossi M, Morrison M, Holtmann G, Kelly JT, Shanahan ER, Staudacher HM, Campbell KL. Dietary fiber intervention on gut microbiota composition in healthy adults: a systematic review and meta-analysis. Am J Clin Nutr. 2018 Jun 1;107(6):965-983. doi: 10.1093/ajcn/nqy041. PMID 29757343
- [Background] Spoelder M, Koopmans L, Hartman YAW, Bongers CCWG, Schoofs MCA, Eijsvogels TMH, Hopman MTE. Supplementation with Whey Protein, but Not Pea Protein, Reduces Muscle Damage Following Long-Distance Walking in Older Adults. Nutrients. 2023 Jan 10;15(2):342. doi: 10.3390/nu15020342. PMID 36678213
- [Background] Ticinesi A, Nouvenne A, Cerundolo N, Catania P, Prati B, Tana C, Meschi T. Gut Microbiota, Muscle Mass and Function in Aging: A Focus on Physical Frailty and Sarcopenia. Nutrients. 2019 Jul 17;11(7):1633. doi: 10.3390/nu11071633. PMID 31319564
- [Background] Villani A, Wright H, Slater G, Buckley J. A randomised controlled intervention study investigating the efficacy of carotenoid-rich fruits and vegetables and extra-virgin olive oil on attenuating sarcopenic symptomology in overweight and obese older adults during energy intake restriction: protocol paper. BMC Geriatr. 2018 Jan 5;18(1):2. doi: 10.1186/s12877-017-0700-4. PMID 29304744
- [Background] Visser M, Deeg DJ, Lips P; Longitudinal Aging Study Amsterdam. Low vitamin D and high parathyroid hormone levels as determinants of loss of muscle strength and muscle mass (sarcopenia): the Longitudinal Aging Study Amsterdam. J Clin Endocrinol Metab. 2003 Dec;88(12):5766-72. doi: 10.1210/jc.2003-030604. PMID 14671166
- [Background] Wicherts IS, van Schoor NM, Boeke AJ, Visser M, Deeg DJ, Smit J, Knol DL, Lips P. Vitamin D status predicts physical performance and its decline in older persons. J Clin Endocrinol Metab. 2007 Jun;92(6):2058-65. doi: 10.1210/jc.2006-1525. Epub 2007 Mar 6. PMID 17341569
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- [Background] Wu Q, Xu Z, Huang W, Qi X, Wu J, Du J, Kan J. Effect of high plant protein/peptide nutrition supplementation on knee osteoarthritis in older adults with sarcopenia: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2024 Sep;43(9):2177-2185. doi: 10.1016/j.clnu.2024.07.037. Epub 2024 Aug 6. PMID 39142111
- [Background] Xu ZR, Tan ZJ, Zhang Q, Gui QF, Yang YM. The effectiveness of leucine on muscle protein synthesis, lean body mass and leg lean mass accretion in older people: a systematic review and meta-analysis. Br J Nutr. 2015 Jan 14;113(1):25-34. doi: 10.1017/S0007114514002475. Epub 2014 Sep 19. PMID 25234223
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478